CLINICAL TRIAL: NCT06242730
Title: Doxycycline PEP and 4CMenB as a Comprehensive Prevention Strategy in MSM and TGW at High Risk for Bacterial STIs Within the Swiss HIV Cohort Study
Acronym: DOXY-MEN
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss HIV Cohort Study (Network)
Responsible Party: Sponsor
Other Study IDs: BASEC-Nr. 2023-01057
Record Dates: First submitted 2024-01-09; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Doxycycline STI PEP
Keywords: Docycycline; Postexposure Propylaxis; Bacterial sexaully tarnsmitted diseases; Sexuylly transmitted diseases; People living with HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — STI swabs (urethra, throat, rectal), stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People living with HIV participating in the Swiss HIV Cohort Study on doxycycline STI PEP: The target population for this study are MSM or TGW at high risk for a bacterial STI (≥1 occasional partners within the preceding 6 months) taking teh doxycycline STI PEP

SUMMARY:
The study aims at assessing effectiveness of offering event-driven Doxy PEP and 4CMenB immunization in MSM/TGW at high STI risk. It plans to offer this STI prevention package to all MSM/TGW in the SHCS who are at risk of STI and then comparing 12-months STI incidence between those accepting and those not accepting the prevention package. The proposal further hosts two interesting sub-studies: One assessing potential effect of Doxy PEP on the microbiome and the other one assessing potential impact of Doxy PEP on TP, MG and CT resistance.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years of age

* Participant in the SHCS
* On antiretroviral therapy with suppressed viral load for ≥ 3 months
* MSM or TGW
* ≥ 1 bacterial STI (syphilis, CT, MG, or NG) within the past 3 years and/or reporting condomless sex with ≥ 1 occasional partner within the last 6 months
* Consenting for off-label use of doxycycline as PEP and/or 4CMenB for the prevention of bacterial STIs
* No allergy or intolerance to doxycycline or 4CMenB
* No other contraindication for doxycycline (e. g. co-medication)

Exclusion Criteria:

* Not participating in the SHCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study are MSM or TGW at high risk for a bacterial STI (≥1 occasional partners within the preceding 6 months).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of bacterial STIs | From enrolment until the date of first event, assessed up to 96 weeks
  Overall incidence of bacterial STIs (including syphilis, CT, NG and MG)
Overall prevalence of bacterial STIs | From enrolment to end of study, i.e. up to 96 weeks
  Overall period prevalence of bacterial STIs (including syphilis, CT, NG and MG)
STI incidence by individual infectious agent | From enrolment until the date of first event, assessed up to 96 weeks
  STI incidence by individual infectious agent (syphilis, CT, NG; and MG if it is included in the local multiplex PCR panel)
STI period prevalence by individual infectious agent | From enrolment to end of study, i.e. up to 96 weeks
  STI period prevalence by individual infectious agent (syphilis, CT, NG; and MG if it is included in the local multiplex PCR panel)

SECONDARY OUTCOMES:
Acceptance of the intervention | From enrolment assessed up to 96 weeks
  Web-based online questionnaire on acceptance of the intervention implemented in the SHCS DJANGO tool assessed once for every participant during the whole study period
Safety and adherence | From enrolment assessed up to 96 weeks
  Web-based online questionnaire on safety and adherence of the intervention implemented in the SHCS DJANGO tool, assessed at every SHCS visit (i.e. every six months)
Genotypic resistance testing of STIs | From enrolment assessed up to 96 weeks
  Genotypic resistance testing for STIs either by whole genome sequencing or "SureSelect" approach performed at the time of detection of each STI
Microbiome of the urethra and the rectum | From enrolment assessed up to 96 weeks
  Genotypic resistance testing for STIs either by whole genome sequencing or "SureSelect" approach performed at every SHCS visit (i.e. every six months)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided